CLINICAL TRIAL: NCT06680232
Title: A Phase 1, Open-Label, First-in-Human, Dose Escalation (Part 1) and Expansion (Part 2) Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of PBGENE-HBV in Participants With Chronic Hepatitis B (ELIMINATE-B)
Brief Title: Phase 1 Study to Evaluate Safety and Antiviral Activity of PBGENE-HBV in Adult Patients With Chronic Hepatitis B
Acronym: ELIMINATE-B
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Precision BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBGENE-HBV-01
Record Dates: First submitted 2024-10-24; First posted 2024-11-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: HEPATITIS B CHRONIC
Keywords: HEPATITIS B CHRONIC; Gene Therapy; Gene Editing; PBGENE-HBV
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: Part 1 is to identify a safe and well tolerated dose regimen of PBGENE-HBV Part 2 is an expansion cohort to aid in selecting a dosing regimen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Participants in both Part 1 and 2 will receive a finite course of PBGENE-HBV. (Experimental): All participants will receive a finite course of multiple IV dose administrations of PBGENE-HBV. In Part 1, this will be done in a dose escalation manner which may be evaluated further in a Part 2 expansion cohort.
  Interventions: Biological: PBGENE-HBV

INTERVENTIONS:
Biological: PBGENE-HBV — PBGENE-HBV is an in vivo gene editing intervention based on a novel proprietary ARCUS® platform designed to potentially cure chronic hepatitis B virus (HBV) by eliminating cccDNA, the key source of replicating hepatitis B virus, while also inactivating integrated HBV DNA in hepatocytes.

SUMMARY:
This is a Phase 1, open-label, dose escalation and dose expansion study to evaluate the safety, tolerability, PK, and antiviral activity of PBGENE-HBV in adult participants with chronic hepatitis B.

DETAILED DESCRIPTION:
Refer to key Inclusion and Exclusion criteria.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or women of non-child bearing potential
* BMI 18.0 to 35.0
* Good overall health deemed by the study Investigator
* CHB infection documented at least 12 months prior to screening
* HBeAg-negative CHB
* Must be virologically suppressed on current NA treatment

Key Exclusion Criteria:

* No history of cirrhosis of the liver
* No current infections of Hepatitis A, D, and E, human immunodeficiency virus (type 1 and 2), and no history of or current hepatitis C. In addition, no other active infections deemed clinically relevant.
* No signs of hepatocellular carcinoma
* Not received an organ transplant
* No malignancy within 5 years of screening, except for specific cancers that are cured by surgical resection (e.g., basal cell skin cancer)
* No investigational agent received within 6 months of screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Safety to Assess Treatment-emergent Adverse Events (TEAEs) | 4 weeks after final dose
  Frequency of TEAEs

SECONDARY OUTCOMES:
Additional Safety | 48 weeks
  Frequency and severity of adverse events and changes in physical examinations, vital signs, and safety labs (hematology, chemistry, and urinalysis)
Pharmacokinetics of AUC | 4 weeks
  Total PBGENE-HBV exposure over time
Pharmacokinetics of Cmax | 4 weeks
  Time at which Cmax (maximum peak concentration of PBGENE-HBV) is observed
Pharmacokinetics of Cmin | 4 weeks
  Minimum (or trough) concentration of PBGENE-HBV
Pharmacokinetics of half life (t1/2) | 4 weeks
  Terminal half life
Antiviral Activity of HBsAg and Anti-HBs | 48 weeks
  Changes from baseline in hepatitis B surface antigen (HBsAg) and anti-HBs levels
Antiviral Activity of HBV DNA | 48 weeks
  Changes from baseline of HBV DNA

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Frankel, MD Medical Monitor, Study Director — Precision BioSciences, Inc.
Locations (4):
- Massachusetts General Hospital/Harvard University, Boston, Massachusetts, United States
- Queen Mary Hospital, The University of Hong Kong, Hong Kong, Hong Kong, Hong Kong
- ICS ARENSIA Exploratory Medicine SRL, Chisinau, Moldova
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No